CLINICAL TRIAL: NCT02475018
Title: The Effect of Shuhua Milk Fortified With Plant Sterol Esters on Serum Cholesterol in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YL/CL-004
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-07

CONDITIONS: Hypercholesterolemia
Keywords: Shuhua Milk; plant sterol esters; serum cholesterol; human
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk fortified with plant sterol esters (Experimental): 250mL of Shuhua Milk fortified with plant sterol esters(with plant sterol esters 262mg/100mL) has been taken twice per day. 500mL of Shuhua milk in total has been taken per day during the 60-days intervention.
  Interventions: Dietary Supplement: Milk fortified with plant sterol esters
- Plain milk (Placebo Comparator): 250mL of placebo milk(plain milk) has been taken twice per day. 500mL of plain milk in total has been taken per day during the 60-days intervention.
  Interventions: Dietary Supplement: Plain milk
- No dairy product consumption (No Intervention): Participants have not consumed any dairy product during the 60-days of study period.

INTERVENTIONS:
Dietary Supplement: Milk fortified with plant sterol esters — 250mL of Shuhua milk fortified with plant sterol esters(with plant sterol esters 262mg/100mL) has been taken twice per day. 500mL of Shuhua milk in total has been taken per day during the 60-days intervention.
  Arms: Milk fortified with plant sterol esters
Dietary Supplement: Plain milk — 250mL of placebo milk (plain milk) has been taken twice per day. 500mL of plain milk in total has been taken per day during the 60-days intervention.
  Arms: Plain milk

SUMMARY:
The purpose of this study is to determine whether YiLi Xinhuo Shuhua Milk is effective in reducing the serum cholesterol in human with hypercholesterolemia.

DETAILED DESCRIPTION:
In a randomized, placebo-controlled double-blind mono-centric study,179 subjects with total cholesterol (TC) level above 5.18mmol/L and triglyceride (TG) level lower than 2.25mmol/L were assigned to 500ml of low lactose milk enriched with 1.58g plant sterol esters or 500ml plain milk without plant sterols (placebo) or without any dairy product consumption (control) for 60 days. Subjects were instructed to maintain stable diet pattern and physical activity. Plasma concentrations of TC,TG,LDL cholesterol(LDL-C) and HDL cholesterol(HDL-C) were measured at initial visits, after 30days and after 60 days. The primary measurement was the change in TC. Secondary measurements were changes in TG,LDL-C and HDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-65 yrs;
* Serum TC ≥5.18mmol/L, and TG≤2.25mmol/L;
* Normal blood pressure or able to control blood pressure within normal range;
* Willing to consent to study participation and to comply with study requirements.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Known allergies to dairy and any substance in the study product.For example lactose intolerance;
* Any comorbidity that could,in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes, including but not limited to cardiac disease, hepatic disease, renal disease, hematopoietic system disease and mental disease;
* Recent use (within 2 weeks of screening) of any prescription or OTC medication that affects serum total cholesterol or that may confound study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Total Cholesterol(TC) during and after intervention | Baseline & 1 months & 2 mongths

SECONDARY OUTCOMES:
Change in Triglyceride(TG) during and after intervention | Baseline & 1 months & 2 mongths
Change in LDL-C level during and after intervention | Baseline & 1 months & 2 mongths
Change in HDL-C level during and after intervention | Baseline & 1 months & 2 mongths

CONTACTS AND LOCATIONS:
Overall Officials: Ignatious Szeto, Ph.D, Study Director — Inner Mongolia Yili Industrial Group Co., Ltd; Jing Zhu, Principal Investigator — Beijing Research Institute for Nutrition Resources
Locations (1):
- BaiZhiFang Community Health Service Centre, Beijing, Beijing Municipality, China